CLINICAL TRIAL: NCT06157411
Title: Validation of a Mindful Eating Program Adapted to the French Population Living With Overweight or Obesity
Brief Title: Adapting Mindful Eating Program for French Overweight/Obese Population
Acronym: MIND-EAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL22_0210
Record Dates: First submitted 2023-11-17; First posted 2023-12-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obesity
Keywords: Mindful eating; Mindfulness; Validation program; Mixed methods
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Eating Intervention (AC group) (Experimental): * Mindful eating program: Two sub-groups of 14 participants will follow the program for 8 consecutive weeks.
  * Follow-up group session: The two groups of 14 participants will each attend a follow-up group session.
  * 3 visits with a doctor: The 28 participants will have a pre-intervention visit, a post-intervention visit, and a final visit 3 months after the program.
  * Focus groups: The two groups of 14 participants will be divided into two (N=7, x4) for a focus group session.
  Interventions: Behavioral: Mindful Eating Intervention (AC group)
- Conventional Dietetic Intervention (DC group) (Active Comparator): * Therapeutic education program (ETP): The 28 participants will follow the ETP program "Obesity: living better, balancing my weight".
  * Follow-up group session: The 28 participants will have an individual follow-up session in the form of a final Shared Educational Assessment.
  * 3 visits with a doctor: The 28 participants will have a pre-intervention visit, a post-intervention visit, and a final visit 3 months after the program.
  Interventions: Behavioral: Conventional Dietetic Intervention (DC group)

INTERVENTIONS:
Behavioral: Mindful Eating Intervention (AC group) — Screening visit: Patients will meet with a doctor, a dietician, a teacher of adapted physical activity or a psychologist.
  Visit 0: Following 24 to 72 hours of reflection, the investigator will confirm the patient's understanding of the study, and those expressing verbal willingness will be randomized into the two groups.
  Visit 1: Participants will be weighed and required to fill out eight questionnaires on a secure platform.
  Mindful eating program: group sessions one evening a week (8x2h) and home exercises (30 min/day).
  Visit 2: visit identical to visit 1
  Follow-up group session: To assess each person's progress according to their needs, resources, difficulties, life plans, and initial expectations.
  Visit 3: visit identical to visit 1
  Focus groups: Each participant will be asked to describe the program and talk about their perceptions and feelings, as well as the potential changes in behavior they have observed in their daily life.
  Arms: Mindful Eating Intervention (AC group)
Behavioral: Conventional Dietetic Intervention (DC group) — Screening visit: Patients will meet with a doctor, a dietician, a teacher of adapted physical activity or a psychologist.
  Visit 0: Following 24 to 72 hours of reflection, the investigator will confirm the patient's understanding of the study, and those expressing verbal willingness will be randomized into the two groups.
  Visit 1: Participants will be weighed and required to fill out eight questionnaires on a secure platform.
  Visit 2: visit identical to visit 1
  Follow-up group session: To assess each person's progress according to their needs, resources, difficulties, life plans, and initial expectations.
  Visit 3: visit identical to visit 1
  Arms: Conventional Dietetic Intervention (DC group)

SUMMARY:
The aim of this project is to validate a new mindful eating programme adapted to the overweight or obese French population. Recognising the importance of diet in the management of chronic diseases, particularly obesity, and the limitations of traditional weight management approaches, the study focuses on the application of mindful eating. The investigators have adapted a model based on an existing eating disorders programme overseas, taking into account feedback from participants in a qualitative study and the scientific literature. The ultimate aim is to test and validate the effectiveness of this new programme in improving the care of overweight or obese French adults, thereby filling a gap in interventions for this population in France.

DETAILED DESCRIPTION:
This research will take the form of a single-center, randomized, two-arm trial comparing a mindful eating intervention (AC group) with a conventional dietary intervention (DC group). The investigators plan to enroll 56 patients who will be randomized to these two groups with stratification based on gender, age (<45, >=45), and BMI (25-30, >30). Randomization will be performed by minimization.

Participants in the AC group (N=28) will follow a program led by an instructor trained in nutrition and mindfulness, incorporating the Alberts program adapted for the overweight or obese population. For 8 consecutive weeks, comprising one 2-hour group session per week at Montpellier University Hospital and individual exercises at home.

Participants in the DC group (N=28) will follow the standard weight management program normally offered by the Nutrition - Diabetes Unit of the Montpellier University Hospital.

This research also includes a qualitative study for the AC group, based on focus groups set up after the end of the mindful eating program.

Participants will be recruited from all consecutive overweight or obese patients attending the Nutrition and Diabetes Unit of the University Hospital of Montpellier who have not yet been enrolled in the therapeutic education program. The unit sees over 1,000 patients a year who meet the criteria for this study.

ELIGIBILITY:
Inclusion Criteria:

* First visit to the Nutrition and Diabetes Unit of Montpellier University Hospital for overweight/obesity
* Adults aged 18 and over, volunteers
* BMI ≥ 25kg/m² and ≤ 50kg/m²
* Provisional verbal consent followed by signed written consent

Exclusion Criteria:

* People who are illiterate or suffer from a major cognitive impairment that prevents them from understanding the study and the mindful eating program
* Pregnant or breast-feeding women
* People who are taking medicines that may have an effect on their weight (especially GLP-1 analogs, neuroleptics, corticosteroids)
* Anyone with a history of bariatric surgery or scheduled bariatric surgery within the next 6 months
* Presence of co-morbidities or severe pathologies (in particular respiratory failure, heart failure, cancer)
* Diagnosis of severe psychiatric disorder (in particular schizophrenia, bipolar disorder), depressive syndrome, or suicidal behavior in the past year
* People suffering from genetic or syndromic obesity
* Lack of Internet access
* Person currently participating in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Variation in the level of mindful eating. | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by the Mind-Eat Scale questionnaire. The Mind-Eat Scale is the first questionnaire to provide a total score of the level of mindful eating and is available in French. This questionnaire was developed and validated as part of the Mind-eat project led by our research team, and the corresponding scientific publication is currently being published.

SECONDARY OUTCOMES:
Variation in anxiety and depression levels. | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by the Hospital Anxiety and Depression scale (HAD) questionnaire. The HAD scale is a screening instrument for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven to depression (total D), giving two scores (maximum score for each = 21).
  A score of 0 to 7 means: no symptoms A score between 8 and 10 means: doubtful symptomatology A score of 11 to 21 means: definite symptomatology The higher the score, the more stress and depression are present.
Variation in the level of intuitive eating. | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by the IES-2-French version questionnaire.
Variation in the level of compulsive eating. | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by the BES-French version questionnaire.
Variation in the level of mindfulness. | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by the FFMQ-French version questionnaire.
Variation in eating behavior. | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by the DEBQ-French version questionnaire.
Variation in physical activity levels. | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by the Ricci-Gagnon metric questionnaire.
Variation in stress levels. | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by the PSS-French version questionnaire.
Gross weight loss (kg) | Assess at visit 1 (10 days before program start), visit 2 (7 days after program end) and visit 3 (3 months after program end).
  It will be measured by a doctor from the Nutrition-Diabetes Department of the Montpellier University Hospital.

OTHER OUTCOMES:
Impact of the program on participants' lives | 3 months and 3 weeks after the end of the program
  The focus groups will highlight changes in behavior, points of view, positive or negative experiences, and/or suggestions for improving the program.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Avignon, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Antoine Avignon, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Van Beekum M, Shankland R, Rodhain A, Robert M, Marchand C, Herry A, Prioux C, Touvier M, Barday M, Turgon R, Avignon A, Leys C, Peneau S. Development and validation of the mindful eating scale (mind-eat scale) in a general population. Appetite. 2024 Aug 1;199:107398. doi: 10.1016/j.appet.2024.107398. Epub 2024 May 6. PMID 38710449
- [Result] Paolassini-Guesnier P, Van Beekum M, Kesse-Guyot E, Baudry J, Shankland R, Rodhain A, Bellicha A, Leys C, Hercberg S, Touvier M, Alles B, Peneau S. Mindful eating is associated with a healthier plant-based diet in the NutriNet-Sante study. Sci Rep. 2025 Jun 6;15(1):19928. doi: 10.1038/s41598-025-02195-5. PMID 40481021
- [Result] Paolassini-Guesnier P, Van Beekum M, Kesse-Guyot E, Baudry J, Srour B, Bellicha A, Shankland R, Rodhain A, Leys C, Hercberg S, Touvier M, Alles B, Peneau S. Mindful eating is associated with a better diet quality in the NutriNet-Sante study. Appetite. 2025 Feb 1;206:107797. doi: 10.1016/j.appet.2024.107797. Epub 2024 Dec 3. PMID 39638150